CLINICAL TRIAL: NCT06249503
Title: Ultrasound Guided Activated and Non-activated Platelet Rich Plasma Injection Versus Hydro Dissection for Treatment of Carpal Tunnel Syndrome
Brief Title: Ultrasound Guided Activated and Non Activated Platelet Rich Plasma Injection Versus Hydro Dissection by Steroids.
Acronym: PRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 154 2022
Record Dates: First submitted 2023-05-12; First posted 2024-02-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome; Compare Steroids Versus PRP in Dissection of Median Nerve by Ultrasound
Keywords: PRP, CTS
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Activated PRP (Active Comparator): PRP is activated by adding 200μl of 0.025 calcium chloride and used in hydrodissection.
  Interventions: Drug: platelet rich plasma
- Non-Activated PRP (Active Comparator): PRP is used directly in hydrodissection.
  Interventions: Drug: platelet rich plasma
- Steroid group (Active Comparator): Hydro dissection using a combination of steroid (Triamcinolone 40mg), local anesthetics and dextrose.
  Interventions: Drug: platelet rich plasma

INTERVENTIONS:
Drug: platelet rich plasma — The patients hand will be facing upwards and slightly extended, the Median nerve will be identified at the inlet of the carpal tunnel. Ultrasound guided injection will be done with the use of the ulnar in-plane technique. with a 25-gage needle will be introduced from the ulnar side of the wrist between carpal tunnel and median nerve.
  Other Names: PRP; steroids

SUMMARY:
PRP represents a promising, nonsurgical option for patients with carpal tunnel syndrome (CTS) with improvement in symptoms compared to placebo, conservative treatment, and local corticosteroid injections at 3-months postintervention. However, the lack of significant long-term results in pain and function demands the presence of future studies to further determine the long-term effect on a large group of homogeneous patients. More over to determine the clinical indications, effect on differing CTS severities, and the effects of preparation, concentration of the platelets and methods of activation of PRP

DETAILED DESCRIPTION:
1. The patients are blinded to the type of drug and the researchers are blinded to the randomization. Randomization will be done using a research randomization program (http://www.randomizer.org)
2. Patients will be randomly divided into three groups; each consists of 30 patients. Group 1 will include patients subjected to ultrasound guided activated PRP injection, group 2 will include patients subjected to ultrasound guided non-activated PRP injection, and group 3 patients will be subjected to ultrasound guided hydro dissection using a combination of steroid (Triamcinolone 40mg), LA (local anesthesia) and dextrose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate idiopathic Carpal Tunnel Syndrome with clinical manifestations, diagnosed by electrophysiological study and ultrasound. CTS grading will be performed on basis of an electrophysiological study following Stevens classification (Stevens; 1997).

  * Early CTS: abnormal findings only in both comparative studies (≥0.5ms difference in peak latency)
  * Mild CTS: abnormal median sensory study (peak latency ≥3.5ms)
  * Moderate CTS: abnormal median sensory study and prolonged median distal motor latency (onset latency ≥4.5ms)
  * Sever CTS: any of the above mentioned abnormalities together with the evidence of axonal loss either by absent median sensory response, low amplitude, or absent median motor response (<2µV)

Exclusion Criteria:

* • Patients suffering from diabetes, hypothyroidism, rheumatoid arthritis, , cervical radiculopathy, polyneuropathy, brachial plexopathy, traumatic nerve injury, thoracic outlet syndrome, coagulopathy

  * Pregnancy
  * Previous corticosteroid injection into the carpal tunnel.
  * Previous carpal tunnel decompressive surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Pain visual analogue scale | 2 weeks,1,3 and 6 months
  Ruler with number on it and the scale by measuring the distance in millimeter from 0 to 10 where is 0 means no pain and 10 means sever disabling pain and in between the different degrees of pain

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | 2 weeks, 1,3 and 6 months
  questionnaire formed of 11 questions each question give grading from 1 to 5 where is 1 means normal and 5 means sever pain and in between different grades

OTHER OUTCOMES:
cross sectional area | 3 months
  change of cross sectional area of median nerve when measuring cross sectional area in millimeter by ultrasound
Nerve conduction study for median nerve | 3 months
  distal Latency in milliseconds of motor and sensory fibers of median nerve

CONTACTS AND LOCATIONS:
Overall Officials: Mona S Kamel, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No